CLINICAL TRIAL: NCT06931522
Title: Effects of Mat and Reformer Pilates Training on Postural Adjustments, Balance, and Walking in Patients With Multiple Sclerosis
Brief Title: Effects of Mat and Reformer Pilates in Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Cagla Ozkul, PhD, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023 - 960
Record Dates: First submitted 2025-03-21; First posted 2025-04-17 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; balance; Pilates; gait
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mat Pilates (Experimental): In Mat Pilates training, exercise balls and elastic bands will be used. The exercises will be done with 10 repetitions for the first 4 weeks, and with 20 repetitions for the last 4 weeks. The difficulty level of the exercises will be increased in the following weeks according to the patient's condition.
  Interventions: Other: Mat Pilates
- Reformer Pilates (Experimental): In the Reformer Pilates group, the difficulty level of the exercises will be provided by different positions, and the springs' resistance will be increased.
  Interventions: Other: Reformer Pilates
- Control group (No Intervention): The control group will perform the relaxing exercise at home.

INTERVENTIONS:
Other: Mat Pilates — In Mat Pilates training, exercise balls and elastic bands will be used. The exercises will be done with 10 repetitions for the first 4 weeks, and with 20 repetitions for the last 4 weeks. The difficulty level of the exercises will be increased in the following weeks according to the patient's condition.
  Arms: Mat Pilates
Other: Reformer Pilates — In the Reformer Pilates group, the difficulty level of the exercises will be provided by different positions, and the springs' resistance will be increased.
  Arms: Reformer Pilates

SUMMARY:
Our study aims to investigate the effects of core stability-based Mat Pilates and Equipment-Based Pilates training on anticipatory postural adjustments (APA), balance, and gait in individuals with Multiple Sclerosis (MS). Participants diagnosed with MS will be randomly assigned to Mat Pilates, Equipment-Based Pilates, or a control group. Both Pilates programs will be conducted twice a week for eight weeks.

Assessments will be conducted before and after the training period. Anticipatory postural adjustments (APA) will be evaluated using electromyography (EMG) electrodes placed on the Erector Spinae and Tibialis Anterior muscles while participants take a step. Biomechanical responses related to APAs, specifically center of pressure displacement, will be measured using a force platform (Biodex® BioSway).

Core endurance will be assessed using the lateral bridge test, Modified Biering-Sorensen test, trunk flexion test, and prone bridge test, while core strength will be evaluated through sit-ups and push-ups. Balance will be measured using posturography. The Activities-Specific Balance Confidence (ABC) Scale will assess confidence in performing daily activities requiring balance. Functional mobility will be evaluated using the Timed Up and Go (TUG) test. Spatiotemporal gait parameters and variability will be analyzed with the BTS® G-WALK system. The Multiple Sclerosis Quality of Life Questionnaire (MSQOL-54) will assess quality of life.

This study is unique in that, unlike previous Pilates studies, it will be the first to examine the effects of different Pilates methods on APAs, which are crucial for both locomotor activities and postural stability in individuals with MS. Additionally, it will be the first study to evaluate two commonly used Pilates techniques in terms of their impact on balance and gait.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis by a specialist physician
* Having a disability level between 0-4.5 according to the Expanded Disability Status Scale (EDSS)
* Being between the ages of 18-65
* Not having had an attack in the last 3 months
* Mini-Mental Test score > 25

Exclusion Criteria:

* Having another neurological disorder
* Having orthopedic, cardiovascular, and pulmonary problems that may affect the research results
* Having vision, hearing, and perception problems
* Having a disease that may affect the immune system, such as infection, cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Anticipatory postural adjustments (APA) | 8 weeks
  Measurement Tool: Biodex-BioSway™ Portable Balance System
  Parameters Assessed: Maximum posterior displacement (cm), maximum lateral displacement (cm)
  Procedure: Participants will take a step following an auditory cue. The magnitude, duration, and latency of medio-lateral and anterior-posterior APAs, as well as the magnitude and speed of the first step, will be recorded separately.
Neuromuscular activation | 8 weeks
  Measurement Tool: Wireless surface EMG sensors
  Muscles Assessed: Erector spinae (µV), Tibialis anterior (µV)
  Procedure: EMG amplitude will be recorded at the onset of APAs, following SENIAM project (Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles) guideline.
Core stability | 8 weeks
  Core stability will be evaluated in terms of endurance and strength. Core endurance will be measured using the McGill Protocol, which includes the Modified Biering-Sorensen trunk extension test, lateral bridge test, trunk flexion test, and prone bridge test. The results will be recorded in seconds. Core strength will be assessed using sit-ups and modified push-ups, where participants will be asked to complete as many repetitions as possible within 30 seconds.
Postural stability | 8 weeks
  Measurement Tool: Portable Balance System
  Parameters Assessed:
  Total stability index
  Anterior-posterior stability index Medio-lateral stability index
  Procedure: Tests performed for 30 seconds (both feet stance) and 10 seconds (single leg stance), repeated three times. Average values will be reported.
Gait kinematics | 8 weeks
  Measurement Tool: BTS G-WALK sensor system
  Parameters Assessed:
  Walking speed (m/s)
  Cadence (steps/min)
  Step length (m)
  Step time (s)
  Stance time (s)
  Swing time (s)
  Double support time (s)
  Single support time (%)
  Pelvic angle changes (degrees)
  Procedure: Participants will walk naturally over a 7-meter course while spatiotemporal parameters are recorded.

SECONDARY OUTCOMES:
Balance Confidence | 8 weeks
  The Activities-Specific Balance Confidence (ABC) Scale will be used to assess participants' perceived balance confidence in 16 daily activities, scored from 0% (completely unconfident) to 100% (completely confident). Lower scores indicate a higher risk of balance impairment and falls.
Mobility | 8 weeks
  Functional mobility will be evaluated using the Timed Up and Go (TUG) test. Participants will be asked to stand up from a chair, walk 3 meters, turn around, return, and sit back down. The test will begin with a verbal "go" command, and the completion time will be recorded in seconds using a stopwatch.
Fatigue severity | 8 weeks
  Fatigue levels will be assessed using the Fatigue Severity Scale (FSS), a 9-item scale where each item is scored from 1 to 7. A total score of 28 or higher indicates severe fatigue, making it particularly useful for individuals with Multiple Sclerosis (MS).
Quality of life | 8 weeks
  Quality of life will be evaluated using the Multiple Sclerosis Quality of Life-54 (MSQOL-54) questionnaire. This 54-item instrument generates 12 subscales along with two summary scores, and two additional single-item measures. The subscales are: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function. The summary scores are the physical health composite summary and the mental health composite summary. The single item measures are satisfaction with sexual function and change in health. This questionnaire, which has been validated in Turkish, will offer a comprehensive assessment of the quality of life in individuals with MS.

CONTACTS AND LOCATIONS:
Overall Officials: Cagla Ozkul, PhD, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez-Fuentes G, Silveira-Pereira L, Ferradans-Rodriguez P, Campo-Prieto P. Therapeutic Effects of the Pilates Method in Patients with Multiple Sclerosis: A Systematic Review. J Clin Med. 2022 Jan 28;11(3):683. doi: 10.3390/jcm11030683. PMID 35160134
- [Background] Massot C, Simoneau-Buessinger E, Agnani O, Donze C, Leteneur S. Anticipatory postural adjustment during gait initiation in multiple sclerosis patients: A systematic review. Gait Posture. 2019 Sep;73:180-188. doi: 10.1016/j.gaitpost.2019.07.253. Epub 2019 Jul 19. PMID 31344607
- [Background] Sever J, Babic J, Kozinc Z, Sarabon N. Postural Responses to Sudden Horizontal Perturbations in Tai Chi Practitioners. Int J Environ Res Public Health. 2021 Mar 7;18(5):2692. doi: 10.3390/ijerph18052692. PMID 33800052
- [Background] Bulguroglu I, Guclu-Gunduz A, Yazici G, Ozkul C, Irkec C, Nazliel B, Batur-Caglayan HZ. The effects of Mat Pilates and Reformer Pilates in patients with Multiple Sclerosis: A randomized controlled study. NeuroRehabilitation. 2017;41(2):413-422. doi: 10.3233/NRE-162121. PMID 28946576